CLINICAL TRIAL: NCT07405112
Title: Impact of Curve Magnitude (Cobb Angle) on Pain Severity and Body Image Perception in Adolescent Idiopathic Scoliosis
Brief Title: Impact of Curve Magnitude on Pain and Body Image in Patients With Adolescents Idiopathic Scoliosis
Acronym: AIS
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Pelin Kacar Yüncü, Principal Investigator, Antalya Training and Research Hospital
Other Study IDs: 2024-090
Record Dates: First submitted 2026-01-29; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Adolescent Idiopathic Scoliosis (AIS); Back Pain; Back Pain Lower Back; Body Image; Pain Severity; Radiographic Study; Scoliosis; SRS
Keywords: Adolescent idiopathic scoliosis; Back pain; lower back pain; Pain severity; Cobb angle; Curve severity; Trunk asymmetry; Radiographic parameters; body image
MeSH Terms: conditions — Back Pain; Low Back Pain; Pain; Scoliosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Low AIS: In this group participants will be patients diagnosed with adolescent idiopathic scoliosis who have a coronal plane Cobb angle of less than 20°, measured on standing posteroanterior spinal radiographs using the Cobb method. This group represents individuals with mild scoliosis.
- Moderate AIS: Participants in this group will be patients diagnosed with adolescent idiopathic scoliosis who have a coronal plane Cobb angle between 21° and 35°, measured on standing posteroanterior spinal radiographs using the Cobb method. This group represents individuals with moderate scoliosis.
- Moderate-to-Severe AIS: Participants in this group will be patients diagnosed with adolescent idiopathic scoliosis who have a coronal plane Cobb angle between 36° and 40°, measured on standing posteroanterior spinal radiographs using the Cobb method. This group represents individuals with moderate-to-severe scoliosis.

SUMMARY:
Adolescent idiopathic scoliosis (AIS) is a three-dimensional spinal deformity characterized by lateral curvature and rotation of the spine. The Cobb angle is the most widely used measurement to quantify the magnitude of spinal deformities. According to the Cobb method, curvatures less than 10 degrees are considered normal spinal asymmetry, whereas curvatures greater than 10 degrees are defined as scoliosis. Based on the coronal Cobb angle, scoliosis is classified as mild (<20°), moderate (21-35°), moderate-to-severe (36-40°), severe (41-50°), severe-to-very severe (51-55°), and very severe (>65°).

AIS occurs in adolescents aged 10-18 years. Although back and low back pain are frequently reported in individuals with AIS, the relationship between curve severity, pain, and body image perception has not been fully elucidated. Furthermore, it remains unclear whether AIS leads to disability or functional limitations, and whether spinal curve severity influences pain intensity. Therefore, further research is required to clarify these issues.

Accordingly, a cross-sectional observational study was designed involving individuals diagnosed with AIS. Participants aged 10-18 years who were diagnosed with AIS and presented to the Scoliosis Clinic of the Physical Medicine and Rehabilitation Department at the University of Health Sciences Antalya Training and Research Hospital will be included. Participants must have no additional comorbid diseases and must voluntarily agree to participate in the study.

Participants will be divided into three groups according to curve severity measured by Cobb angle: Group I (mild, <20°), Group II (moderate, 21-35°), and Group III (moderate-to-severe, 36-40°). Medical history, neurological and physical examinations, and radiological measurements will be performed. Pain will be assessed using the pain-related domain of the Scoliosis Research Society-22 (SRS-22) questionnaire based on participant responses. Body image perception will be evaluated using the Turkish version of the Spinal Appearance Questionnaire (TR-SAQ), completed independently by both participants and evaluators.

Intergroup comparisons will be conducted to evaluate the effects of curve severity on pain and body image perception, and to determine the statistical significance of these associations.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) is considered a risk factor for back and low back pain. Epidemiological studies have shown that, compared with healthy controls, individuals with AIS experience back and/or low back pain more frequently, with greater severity and longer duration, with reported prevalence rates ranging from 23% to 85%. However, the presence, clinical relevance, and determinants of pain in AIS remain controversial. In a systematic review including 15 studies, although 81% of patients with AIS reported severe pain, only 5% of these cases were considered clinically significant. In a prospective study using the Scoliosis Research Society-22 Revised (SRS-22R) questionnaire, no difference in preoperative coronal curve magnitude was observed between patients with and without pain. Another retrospective study reported that patients with thoracic curves experienced more pain compared with those with lumbar curves. Retrospective studies have demonstrated that the lifetime prevalence of back pain is approximately 47% in individuals with AIS and 40% in healthy individuals. However, these studies were limited by unclear definitions of back pain and inconsistent documentation in medical records. In a retrospective study with a 50-year follow-up, individuals with AIS were reported to develop back and/or low back pain regardless of curve magnitude or localization, experiencing more chronic pain and more severe and longer-lasting acute pain than controls. In that study, pain history was not associated with curve severity, and functional capacity in daily and occupational activities was comparable to that of healthy individuals. In another retrospective study, no clear explanatory relationship between spinal deformity and pain was identified, which was attributed to limitations in retrospective pain assessment. Pain intensity and its relationship with activity or rest were not evaluated. Additionally, due to limited assessment of sagittal spinopelvic parameters, the potential effects of sagittal alignment variables, such as sagittal vertical axis or pelvic incidence, were not analyzed. Evidence regarding curve-specific radiological parameters and their relationship with subjective pain scores in AIS remains insufficient. In a study involving surgically indicated AIS patients, lumbar curve magnitude was associated with pain; however, no significant differences were observed when curve type or sagittal characteristics were compared. Although back and low back pain are common in AIS, some studies suggest that pain does not necessarily lead to disability or functional impairment and that curve magnitude may not influence pain severity. Conversely, other reports indicate that increasing curve magnitude may be associated with greater pain, cosmetic deformity, and subjective respiratory discomfort. Overall, the literature lacks consistency regarding pain characteristics, including intensity, duration, localization, relationship with activity, and aggravating or relieving factors. Prospective studies addressing these factors remain limited, and no clear consensus exists regarding the direct effect of curve magnitude or location on pain in AIS. To better understand the burden of pain in AIS and to facilitate effective pain management, systematic assessment of back and low back pain is required, taking into account the multifactorial nature of pain and potential contributing factors. Therefore, a cross-sectional observational study was designed to evaluate the effects of spinal curve severity on pain and body image perception in patients aged 10-18 years diagnosed with AIS. Participants will be recruited from individuals aged 10-18 years diagnosed with AIS who present to the Scoliosis Outpatient Clinic of the Physical Medicine and Rehabilitation Department at Antalya Training and Research Hospital. Individuals with additional comorbidities will be excluded. Participation will be voluntary. Participants will be categorized into three groups based on radiographic Cobb angle measurements: Group I (mild, <20°), Group II (moderate, 21-35°), and Group III (moderate-to-severe, 36-40°). Evaluations will include medical history, physical examination, radiological measurements, structured questionnaires, the pain domain of the Scoliosis Research Society-22 (SRS-22), and the Turkish version of the Spinal Appearance Questionnaire (TR-SAQ). Pain severity will be assessed using the SRS-22 pain domain and the Numerical Rating Scale (NRS). Body image perception will be evaluated using the TR-SAQ. Radiological assessment will be performed subsequently. Standing posteroanterior and lateral spine radiographs will be obtained using a detector measuring 350 × 430 mm, with a source-to-image distance of 2 meters. Images will be acquired with participants standing upright, knees extended, feet shoulder-width apart, and head facing forward. Cobb angles will be measured on standing posteroanterior radiographs, and vertebral rotation will be assessed using the Nash-Moe method. Radiographic measurements will be performed independently by two assessors blinded to clinical data. If the difference between measurements is ≤5°, the mean value will be used; if the difference exceeds 5°, a consensus measurement will be determined. Participants presenting with pain and suspected pathology other than AIS on physical examination will undergo further imaging and laboratory evaluation, and those with additional pathology will be excluded. The study hypotheses are as follows: Pain prevalence increases with increasing curve severity. Pain intensity increases with increasing curve severity. Pain is more frequent in lumbar curves. Vertebral rotation is associated with pain severity. Body image perception worsens with increasing curve severity. A moderate correlation exists between patient-reported and evaluator-assessed body image perception. Sample size was calculated using G*Power version 3.1.9.4 with an effect size of 0.6, statistical power of 90%, two degrees of freedom, and a significance level of 0.05, yielding a required sample size of 66 participants. Allowing for a potential 10% data loss, the final sample size was set at 72 participants. Statistical analyses will be conducted using SPSS version 25.0 (IBM Corp., Armonk, NY, USA). Descriptive statistics will be presented as frequency, percentage, mean, standard deviation, median, minimum, maximum, and interquartile range. Normality will be assessed using the Kolmogorov-Smirnov test, and homogeneity of variance using the Levene test. Group comparisons will be performed using one-way ANOVA or Kruskal-Wallis tests with appropriate post hoc analyses. Categorical variables will be analyzed using Pearson chi-square or Fisher's exact tests. Correlations will be evaluated using Pearson or Spearman correlation coefficients. A p value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation
* Presence of adolescent idiopathic scoliosis (AIS)
* Age between 10 and 18 years
* Cobb angle ≥ 10°

Exclusion Criteria:

* History of spinal or other joint/bone surgery
* Age ≥19 years or ≤9 years
* Presence of spinal or costal deformities other than adolescent idiopathic scoliosis (AIS)
* History of spinal trauma within the past 1 year
* Intellectual disability
* Presence of systemic diseases (rheumatologic, inflammatory, oncologic, - cardiac, respiratory, or neurological disorders)
* Cobb angle > 40°

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will include adolescents aged 10-18 years diagnosed with adolescent idiopathic scoliosis (AIS) who present to the Scoliosis Outpatient Clinic of the Physical Medicine and Rehabilitation Department at Antalya Training and Research Hospital, are able to provide reliable responses, and volunteer to participate.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-11-27 (Actual); Study Completion 2025-11-27 (Actual)

PRIMARY OUTCOMES:
Pain severity assessed by Scoliosis Research Society-22 (SRS-22) Pain Domain | At baseline (single assessment at study enrollment)
  Pain severity was assessed using the pain-related domain of the Scoliosis Research Society-22 (SRS-22) questionnaire.
  The SRS-22 Pain Domain consists of multiple items evaluating pain frequency, pain intensity, and pain-related functional limitations associated with scoliosis.
  Each item is scored on a 5-point Likert scale, with possible scores ranging from 1 to 5.
  The domain score is calculated as the mean of the item scores. Minimum score: 1; Maximum score: 5. Higher scores indicate less pain and better pain-related quality of life, whereas lower scores indicate more severe pain.
Pain severity assessed by Numerical Rating Scale (NRS) | Baseline (cross-sectional assessment)
  Pain intensity was assessed using the Numerical Rating Scale (NRS). The Numerical Rating Scale is a unidimensional patient-reported measure of pain intensity.
  Participants are asked to rate their current back and/or low back pain on an 11-point scale.
  Minimum score: 0 ("no pain"); Maximum score: 10 ("worst pain imaginable"). Higher scores indicate greater pain intensity, whereas lower scores indicate less pain.

SECONDARY OUTCOMES:
Body Image perception assessed by Turkish version of the Spinal Appearance Questionnaire (TR-SAQ) | At baseline (single assessment at study enrollment)
  Body image perception will be assessed using the Turkish version of the Spinal Appearance Questionnaire (TR-SAQ). The questionnaire evaluates the individual's perception of body appearance related to spinal deformity. TR-SAQ consists of 10 pictorial items assessing patients' subjective perception of spinal deformity. Each item is scored on a 5-point scale ranging from 1 (least severe deformity) to 5 (most severe deformity). The total Appearance score ranges from 10 to 50, with higher scores indicating worse perceived spinal appearance.

CONTACTS AND LOCATIONS:
Overall Officials: NACİYE F TORAMAN, MD, Principal Investigator — Antalya Training and Research Hospital, Physical Medicine and Rehabilitation Department
Locations (1):
- Antalya Training and Research Hospital, Antalya, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available outside the study team.

REFERENCES:
- [Background] Teles AR, St-Georges M, Abduljabbar F, Simoes L, Jiang F, Saran N, Ouellet JA, Ferland CE. Back pain in adolescents with idiopathic scoliosis: the contribution of morphological and psychological factors. Eur Spine J. 2020 Aug;29(8):1959-1971. doi: 10.1007/s00586-020-06489-2. Epub 2020 Jun 9. PMID 32519028
- [Background] Huskisson EC, Hart FD. Severe, unusual, and recurrent infections in rheumatoid arthritis. Ann Rheum Dis. 1972 Mar;31(2):118-21. doi: 10.1136/ard.31.2.118. No abstract available. PMID 5016859
- [Background] Wong AYL, Samartzis D, Cheung PWH, Cheung JPY. How Common Is Back Pain and What Biopsychosocial Factors Are Associated With Back Pain in Patients With Adolescent Idiopathic Scoliosis? Clin Orthop Relat Res. 2019 Apr;477(4):676-686. doi: 10.1097/CORR.0000000000000569. PMID 30516661